CLINICAL TRIAL: NCT03799614
Title: Vibration Impact on Parkinson's Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM20012404
Record Dates: First submitted 2018-12-19; First posted 2019-01-10 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Lower dose vibration (Experimental): RMBand lower dose vibration
  Interventions: Device: RMBand lower dose
- Higher dose vibration (Experimental): RMBand higher dose vibration
  Interventions: Device: RMBand higher dose

INTERVENTIONS:
Device: RMBand lower dose — Light-weight portable device that delivers low dose vibration to the arm
  Arms: Lower dose vibration
Device: RMBand higher dose — Light-weight portable device that delivers higher dose vibration to the arm
  Arms: Higher dose vibration

SUMMARY:
The primary purpose of this study is to test the safety, tolerability and efficacy of vibration (delivered by an experimental device called RMBand that is worn on the subject's arm) on parkinsonian tremor. The RMBand was developed by Resonate Forward, LLC (RF). This RMBand is designed to administer a vibration to the wearer to decrease or stop tremor in persons with Parkinson's disease (PD).

DETAILED DESCRIPTION:
Participation will be completed in one visit at VCU Parkinson's and Movement Disorders Center. A baseline Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) will be taken prior to vibration therapy. The RMBand (experimental device) will be placed on the arm of the participant to provide the vibration therapy. The MDS-UPDRS Part III will be repeated both during and after the therapy. Participants will be asked to provide feedback about the device, the therapy session and how they are feeling.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease (PD) as diagnosed by a movement disorder specialist
* Tremor caused by their Parkinson's disease
* Ability to provide informed consent

Exclusion Criteria:

* Known diagnosis of Parkinson Plus Syndrome
* Dementia
* Other known non-PD cause of tremor
* Other known non-PD cause of limb dysfunction
* Presence of implantable cardiac device, severe neuropathy or sensory loss that would prevent perception of vibration stimulus
* Non-English speaker
* Prisoners
* Pregnant women

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Pretzer-Aboff, PhD, RN, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose Vibration: RMBand lower dose vibration
  RMBand lower dose: Light-weight portable device that delivers low dose vibration to the arm
- High Dose Vibration: RMBand higher dose vibration
  RMBand higher dose: Light-weight portable device that delivers higher dose vibration to the arm
Period: Overall Study
Arm/Group | Low Dose Vibration | High Dose Vibration
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lower Dose Vibration | Higher Dose Vibration | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (6.7) | 67.6 (8.4) | 67.4 (7.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 11 | 7 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Clinical Rating Scale for Tremor, total score [Mean (Standard Deviation); unit: units on a scale] | 21.13 (10.69) | 18.07 (5.22) | 19.6 (8.55)
MDS UPDRS II - IV total [Mean (Standard Deviation); unit: units on a scale] — Movement Disorder Society Unified Parkinson Rating Scale, (MDS UPDRS, score for parts II - !V.
  units on a scale | 44.26 (16.41) | 38.47 (14.08) | 41.37 (15.56)

OUTCOME MEASURES:

1. Primary Outcome: Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS)
Description: The "Movement Disorder Society Unified Parkinson Disease Rating Scale" (MDS-UPDRS) Part III, only, will be used at baseline, and repeated during vibration and post vibration data collection times. It is a validated scale administered by a clinician, contains 34 items to score between 0 (normal) and 4 (severe). The score range is 0 - 136. It takes ~ 5 minutes to complete. Lower scores are better. This outcome measure will be used to report a change in PD motor symptoms over time.
Time Frame: This rating scale will be used at baseline, 5 minutes after vibration starts, and 5 minutes after vibration is turned off.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Low Dose Vibration: RMBand low dose vibration
  RMBand: Light-weight portable device that delivers low dose vibration to the arm
- Higher Dose Vibration: RMBand high dose vibration
  RMBand: Light-weight portable device that delivers higher dose vibration to the arm
Arm/Group | Low Dose Vibration | Higher Dose Vibration
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline | 32.67 (12.88) | 27.4 (11.25)
  During vibration treatment | 33.67 (14.31) | 27.33 (11.14)
  Post vibration treatment | 32.67 (13.67) | 28.6 (10.39)

2. Primary Outcome: Clinical Rating for Tremor
Description: Clinical Rating Scale for Tremor (Fahn, Tolosa, & Marin) assesses severity of tremor symptoms. This scale takes 10-minutes, Items 1 - 14 will be used to report average changes in tremor.
  Items are rated on a scale of 0=normal to 4=severely abnormal, total summative score range for items 1- 14 points is 0 - 56. Lower scores are better. Total time to complete the Scale for Tremor assessment is 10 minutes.
Time Frame: Data collection times were baseline, 5 minutes after vibration start (vibration duration was 20 minutes), 5 minutes after vibration was stopped. .
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lower Dose Vibration | Higher Dose Vibration
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline | 15.47 (7.94) | 13.87 (4.03)
  During vibration | 15.87 (8.55) | 13.20 (4.03)
  Post vibration | 14.53 (7.98) | 14.13 (5.63)

3. Primary Outcome: Objective Measurement of Tremor Frequency (Hz)
Description: This is a device that will objectively measure tremors frequency and amplitude pre, during, and post treatment.
Time Frame: Five minutes before vibration is turned on, throughout vibration treatment, and approximately five minutes post treatment.
Measure: Mean (Standard Deviation); unit: hertz
Arm/Group | Low Dose Vibration | Higher Dose Vibration
Number analyzed (Participants) | 15 | 15
hertz
  Baseline | 4.77 (1.57) | 4.51 (1.31)
  During Vibration | 4.79 (1.13) | 3.99 (1.12)
  Post Vibration | 3.36 (0.87) | 4.64 (1.48)

4. Primary Outcome: Objective Measurement of Tremor Amplitude (mm).
Description: This is a device that will objectively measure tremor amplitude pre, during, and post treatment.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Low Dose Vibration Amplitude: RMBand low dose vibration
  RMBand: Light-weight portable device that delivers low dose vibration to the arm,reported in mm.
Arm/Group | Low Dose Vibration Amplitude | Higher Dose Vibration
Number analyzed (Participants) | 15 | 15
millimeters
  Baseline | 0.71 (0.82) | 0.43 (0.41)
  During vibration | 0.76 (0.72) | 0.44 (0.31)
  Post vibration | 0.70 (0.75) | 0.52 (0.47)

ADVERSE EVENTS:
Time Frame: two hours, during time of study activities
Groups:
- Lower Dose Vibration: RMBand lower dose vibration
  RMBand lower dose: Light-weight portable device that delivers low dose vibration (frequency of 80 Hz) to the arm
- Higher Dose Vibration: RMBand higher dose vibration
  RMBand higher dose: Light-weight portable device that delivers higher dose (frequency of 160 Hz) vibration to the arm
Arm/Group | Lower Dose Vibration | Higher Dose Vibration
All-Cause Mortality (participants affected / at risk) | 0/15 | 1/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower Dose Vibration (N=15) | Higher Dose Vibration (N=15)
muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — tightness in muscles in right shoulder and neck

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Informed Consent Form (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT03799614/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT03799614/Prot_SAP_002.pdf